CLINICAL TRIAL: NCT00950560
Title: An Empirical Study of Perceived Hospital Service Quality: A Comparison of Inpatient, Outpatient and Emergence Patient
Status: Completed | Type: Observational
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Institutional Review Board, Taipei Municipal Wan Fang Hospital
Other Study IDs: WanFangH98043
Record Dates: First submitted 2009-07-30; First posted 2009-08-03 (Estimated); Last update posted 2011-04-26 (Estimated); Status verified 2011-04

CONDITIONS: Service Quality; Satisfaction
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- inpatient
- outpatient
- emergency patient

SUMMARY:
The authors employ a questionary approach to understanding the relational among patients' perceptions of inpatient, outpatient and emergency room service and their overall perceptions of service quality, satisfaction with hospital.The questionary was applied in total 300 patients (100 inpatients, 100 outpatients and 100 emergency patients).

ELIGIBILITY:
Inclusion Criteria:

* Patients who want to write our questionary.

Exclusion Criteria:

* Patients who reject to write our questionary.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 100 inpatient 100 outpatient 100 emergency patient
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2009-06; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Chih Wang, MD, Principal Investigator — Taipei Medical University-Wan Fang Hospital
Locations (1):
- Taipei Municipal Wan Fang Hospital, Taipei, Taiwan